CLINICAL TRIAL: NCT04773678
Title: A Multicenter, Randomized, Double-blind, Parallel Group, Placebo-controlled, Efficacy and Safety Study of CBP-201 in Patients With Moderate to Severe Persistent Asthma With Type 2 Inflammation
Brief Title: Efficacy and Safety of CBP-201 in Patients With Moderate to Severe Persistent Asthma With Type 2 Inflammation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Connect Biopharm LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CBP-201-WW002
Record Dates: First submitted 2021-02-24; First posted 2021-02-26 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2022-12

CONDITIONS: Moderate to Severe Persistent Asthma
Keywords: Type 2 inflammation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- CBP-201 Dose 1 (Experimental): CBP-201 Dose 1 subcutaneous (SC) injection.
  Interventions: Drug: CBP-201
- CBP-201 Dose 2 (Experimental): CBP-201 Dose 2 subcutaneous (SC) injection.
  Interventions: Drug: CBP-201
- Placebo (Placebo Comparator): Placebo subcutaneous (SC) injection.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CBP-201 — CBP-201 subcutaneous (SC) injection.
  Other Names: rademikibart
  Arms: CBP-201 Dose 1; CBP-201 Dose 2
Drug: Placebo — Placebo subcutaneous (SC) injection.
  Arms: Placebo

SUMMARY:
This study will evaluate the efficacy, safety of two dose levels of CBP-201 in patients with moderate to severe persistent asthma with Type 2 inflammation.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, parallel group, placebo-controlled study to assess the efficacy and safety of two dose levels of CBP-201 administered to eligible patients with moderate to severe persistent asthma with Type 2 inflammation compared to placebo. CBP-201 is administered as a subcutaneous (SC) injection. The study is divided into a treatment period of 24 weeks and a follow-up period of 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Adult male or female patient aged 18 to 75 years with a physician diagnosis of asthma for a minimum of 12 months, based on the Global Initiative for Asthma (GINA) 2020 Guidelines.
2. Patient is currently receiving treatment with medium to high dose inhaled corticosteroids (ICS) in combination with at least 1 additional reliever/controller for at least 90 days prior to the Screening Visit with a stable dose of ICS at least 28 days prior to the Screening Visit.

   Note:
   * Patients receiving ICS equivalent to ≥ 226 μg fluticasone propionate twice daily or equipotent ICS daily dosage of a maximum of 2000 μg/day fluticasone propionate (or equivalent) in combination with a second reliever/controller (eg, long-acting ß agonist [LABA], leukotriene receptor antagonist [LTRA], long-acting muscarinic antagonist [LAMA], theophylline) are eligible.
   * Patients receiving fluticasone furoate/vilanterol with fluticasone furoate ≥ 200 μg once daily are eligible.
   * Patients receiving budesonide/formoterol with budesonide ≥ 640 μg/day are eligible.
   * Patients requiring a third reliever/controller for their asthma are eligible.
   * Patients requiring maintenance oral corticosteroids (OCS) with a stable dose ≤ 10 mg/day prednisone or equivalent OCS in addition to ICS are eligible; OCS total daily dose must have been stable at least 28 days prior to Screening.
3. Prebronchodilator (trough) forced expiratory volume in the first second of expiration (FEV1) must be 40 to 85% of predicted normal at Screening and predose Baseline.
4. Patients must have ≥ 12% reversibility (and ≥ 200 mL difference) in FEV1 within 15 to 30 minutes after the administration of up to 4 puffs of albuterol/salbutamol at Screening.
5. Blood eosinophil count ≥ 300 cells/μL at Screening.
6. Asthma Control Questionnaire, 6-question (ACQ-6) score ≥ 1.5 at Screening and Baseline.
7. Patient has experienced an asthma exacerbation at least once in the past 12 months, defined here as:

   * Use of physician prescribed systemic corticosteroid [oral or parenteral], or
   * Asthma requiring treatment increase of approximately 4 times the baseline dose of ICS, or
   * Hospitalization or emergency medical care due to asthma.
8. Patient demonstrates acceptable inhaler, peak flow meter, and spirometry techniques during the Screening Period in the opinion of the Investigator.
9. Patient demonstrates at least 70% compliance with usual asthma controller use during Run-in Period, based on their patient diary in the 7 days prior to dosing.
10. Patient demonstrates at least 70% compliance with recording of symptom scores in the patient-reported outcomes (PRO) diary completion during Run-in Period and in their handheld pulmonary function device in the 7 days prior to dosing.
11. Patient is able to understand and willing to sign the informed consent form (ICF).
12. Patient is willing and able to comply with clinic visit schedule and study-related procedures, in the opinion of the Investigator.
13. Male patients and their female partners of child-bearing potential agree to practice adequate and effective forms of contraception through the duration of the study from first dose to 8 weeks after the last dose of study drug.
14. Female patients of childbearing potential who are sexually active with a non-sterilized male partner agree to practice adequate and effective forms of contraception from first dose to 8 weeks after last dose of study drug.

    Exclusion Criteria:

    -

    A patient who meets any of the following criteria will be ineligible to participate in this study:
15. Patient has a current diagnosis of a respiratory disorder other than asthma (eg, active lung infection, chronic obstructive pulmonary disease (COPD), bronchiectasis, pulmonary fibrosis, cystic fibrosis) or other disease associated with elevated peripheral eosinophil counts (eg, allergic bronchopulmonary aspergillosis/mycosis, Churg-Strauss syndrome, hypereosinophilic syndrome).
16. Patient has an acute upper or lower respiratory infection requiring antibiotics or antiviral medication within 30 days prior to the date of informed consent or during the Screening/Run-in Period. Note: Patients must be symptom-free for at least 30 days.
17. Patient experiences ana asthma exacerbation at any time from 1 month prior to the Screening Visit up to and including the Baseline Visit. Exacerbation is defined as:

    * Use of physician prescribed systemic corticosteroid [oral or parenteral], or
    * Asthma requiring treatment increase of approximately 4 times the baseline dose of ICS, or
    * Hospitalization or emergency medical care due to asthma.
18. Current smoker or former smoker with a smoking history of > 10 pack-years. Note: This includes tobacco, marijuana, and vaping products.
19. Patient is undergoing or planning to undergo any elective surgery during the study requiring general anesthesia.
20. Patient has received treatment with any marketed (eg, omalizumab, benralizumab, mepolizumab, reslizumab, dupilumab) or investigational biologic drug for asthma or other diseases within 16 weeks or 5 half-lives prior to randomization, whichever is longer.
21. Patient has received treatment with any investigational nonbiologic drug within 30 days or 5 half-lives prior to randomization, whichever is longer.
22. Patient did not respond favorably to previous dupilumab treatment (e.g. therapy failure or patient experienced an adverse reaction to treatment).
23. Patient has received specific immunotherapy within 3 months prior to randomization. Note: If the patient has received immunotherapy, a 3 month washout period is required following the last dose of immunotherapy.
24. Patient is receiving medications or therapy that are prohibited as concomitant medications.
25. Patient has a known or suspected history of immunosuppression, including history of invasive opportunistic infections, such as aspergillosis, coccidioidomycosis, histoplasmosis, HIV, listeriosis, pneumocystosis, pulmonary non-tuberculosis mycobacteria, or tuberculosis, regardless of infection resolution; or unusually frequent, recurrent, or prolonged infections. Note: Tuberculosis testing will be performed on a country-by-country basis according to local guidelines if required by regulatory authorities or ethics committees (ECs).
26. Patient has positive results at Screening for hepatitis B surface antigen (HBsAg), hepatitis B core antibody (HbsAqHBsAq), or hepatitis C antibody (HbsAqHBsAq) with positive HCV RNA polymerase chain reaction; or positive HIV serology at Screening.
27. Patient has a helminth parasitic infection diagnosed within 24 weeks prior to the date of informed consent that has not been treated with, or has failed to respond to, standard of care therapy.
28. Patient shows evidence of acute or chronic infection requiring treatment with antibacterials, antivirals, antifungals, antiparasitics, or antiprotozoals within 28 days of Screening, or significant viral infections within 28 days of Screening that may not have received antiviral treatment (eg, influenza receiving only symptomatic treatment).
29. Patient receives live (attenuated) vaccinations within 7 days of Screening or plans to receive live (attenuated) vaccinations during the study.
30. Patient has any disorder that is not stable in the opinion of the Investigator and may affect the safety of the patient throughout the study; influence the findings of the studies or their interpretations; or impede the patient's ability to complete the entire duration of study, including, but not limited to, cardiovascular, gastrointestinal, hepatic, renal, neurological, musculoskeletal, infectious, endocrine, metabolic, hematological, psychiatric, or major physical impairment.
31. Patient has any clinically significant abnormal findings in physical examination, vital signs, or safety lab tests during Screening/Run-in Period; or any significant medical history which, in the opinion of the Investigator, may put the patient at risk because of his/her participation in the study, or may influence the results of the study, or the patient's ability to complete entire duration of the study.
32. Patient is being treated with immunosuppressive therapy or biologic therapy for autoimmune disease (eg, rheumatoid arthritis, inflammatory bowel disease, primary biliary cirrhosis, systemic lupus erythematosus, multiple sclerosis).
33. Patient has a prolonged corrected QT (QTc) interval (male > 450 milliseconds, female > 470 milliseconds) or tachyarrhythmia.
34. Patient has any of the following laboratory abnormalities at Screening:

    * Eosinophils > 1500 cells/mmE3 or 1.5*10E9/L
    * Platelets < 100000 cells/mmE3 or 100*10E9/L
    * Creatine phosphokinase (CPK) > 10 times the upper limit of normal (ULN)
    * Alanine aminotransferase (ALT) > 2.5 times the ULN
    * Aspartate aminotransferase (AST) ≥ 2.5 times the ULN
    * Bilirubin > 2 times the ULN.
35. Patient has a history of alcohol or drug abuse within 12 months of Screening.
36. Patient has an allergy to L-histidine, trehalose, or Tween (polysorbate) 80 or a history of a systemic hypersensitivity reaction, other than localized injection site reaction, to any biologic drug.
37. Patient has a history of malignancy within 5 years prior to the Baseline Visit, with the following exceptions: patients with a history of completely treated carcinoma in situ of cervix and nonmetastatic squamous or basal cell carcinoma of the skin are allowed.
38. Female patient is pregnant, planning to become pregnant, or is breastfeeding.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 322 (Actual)
Dates: Start 2021-05-11 (Actual); Primary Completion 2023-08-05 (Actual); Study Completion 2023-09-28 (Actual)

PRIMARY OUTCOMES:
Absolute change in prebronchodilator (trough) forced expiratory volume in the first second of expiration (FEV1) | at Week 12
  Absolute change from Baseline in prebronchodilator (trough) FEV1 at Week 12. To assess the efficacy of CBP-201 (Dose 1 and Dose 2) versus placebo in patients with moderate to severe persistent asthma with type 2 inflammation as measured by lung function improvements.

SECONDARY OUTCOMES:
Absolute change in prebronchodilator (trough) FEV1 | at Weeks 1, 2, 4, 8 and 24
  Absolute change from Baseline in prebronchodilator (trough) FEV1 at Weeks 1, 2, 4, 8 and 24.
Percent change in prebronchodilator (trough) FEV1 | at Weeks 1, 2, 4, 8, 12 and 24
  Percent change from Baseline in prebronchodilator (trough) FEV1 at Weeks 1, 2, 4, 8, 12 and 24.
Change in other lung function measurements | From Baseline to Week 24
  Change from Baseline in other lung function measurements [percentage predicted FEV1, morning and evening peak expiratory flow (PEF)].
Time to severe exacerbation and number of events | From Baseline to Week 24
  Time to severe exacerbation and number of events during the 24 weeks Treatment Period.
Proportion of patients with ≥ 1 asthma exacerbation | From Baseline to Week 24
  Proportion of patients with ≥ 1 asthma exacerbation during the 24 weeks Treatment Period.
Incidence, type and severity of Adverse Event (AE) | From Baseline to Week 32
  Safety endpoints will be summarized by descriptive statistics and narratives where indicated by severity. Safety will be assessed on basis of AEs reported, including SAEs and AESIs.
Pharmacokinetics (Steady-state trough PK profile) | From Baseline to Week 32
  Whole blood for plasma CBP-201 concentrations will be obtained and analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Suzhou Connect, Study Director — Connect Biopharm LLC
Locations (76):
- United States (39):
  - Connect Investigative Site 154, Tucson, Arizona
  - Connect Investigative Site 109, Huntington Beach, California
  - Connect Investigative Site 143, Huntington Beach, California
  - Connect Investigative Site 132, Lancaster, California
  - Connect Investigative Site 125, Mission Viejo, California
  - Connect Investigative Site 103, San Jose, California
  - Connect Investigative Site 161, Hialeah, Florida
  - Connect Investigative Site 114, Hollywood, Florida
  - Connect Investigative Site 142, Leesburg, Florida
  - Connect Investigative Site 104, Miami, Florida
  - Connect Investigative Site 166, Miami, Florida
  - Connect Investigative Site 118, Miami, Florida
  - Connect Investigative Site 162, Miami, Florida
  - Connect Investigative Site 163, Miami, Florida
  - Connect Investigative Site 164, Miami, Florida
  - Connect Investigative Site 105, Miami, Florida
  - Connect Investigative Site 165, Miami Gardens, Florida
  - Connect Investigative Site 110, Miami Lakes, Florida
  - Connect Investigative Site 123, Winter Park, Florida
  - Connect Investigative Site 124, Bangor, Maine
  - Connect Investigative Site 120, White Marsh, Maryland
  - Connect Investigative Site 146, West Bloomfield, Michigan
  - Connect Investigative Site 112, St Louis, Missouri
  - Connect Investigative Site 119, Bellevue, Nebraska
  - Connect Investigative Site 144, North Las Vegas, Nevada
  - Connect Investigative Site 111, Princeton, New Jersey
  - Connect Investigative Site 117, Buffalo, New York
  - Connect Investigative Site 153, New York, New York
  - Connect Investigative Site 122, Winston-Salem, North Carolina
  - Connect Investigative Site 136, Cincinnati, Ohio
  - Connect Investigative Site 147, Toledo, Ohio
  - Connect Investigative Site 107, Edmond, Oklahoma
  - Connect Investigative Site 149, Oklahoma City, Oklahoma
  - Connect Investigative Site 129, Warwick, Rhode Island
  - Connect Investigative Site 116, Austin, Texas
  - Connect Investigative Site 102, Boerne, Texas
  - Connect Investigative Site 121, Dallas, Texas
  - Connect Investigative Site 108, El Paso, Texas
  - Connect Investigative Site 150, Katy, Texas
- China (22):
  - Connect Investigative Site 206, Bengbu, Anhui
  - Connect Investigative Site 201, Beijing, Beijing Municipality
  - Connect Investigative Site 216, Beijing, Beijing Municipality
  - Connect Investigative Site 209, Beijing, Beijing Municipality
  - Connect Investigative Site 215, Beijing, Beijing Municipality
  - Connect Investigative Site 203, Guangzhou, Guangdong
  - Connect Investigative Site 211, Luoyang, Henan
  - Connect Investigative Site 213, Wuhan, Hubei
  - Connect Investigative Site 202, Changsha, Hunan
  - Connect Investigative Site 204, Baotou, Inner Mongolia
  - Connect Investigative Site 214, Baotou, Inner Mongolia
  - Connect Investigative Site 210, Hohhot, Inner Mongolia
  - Connect Investigative Site 205, Wuxi, Jiangsu
  - Connect Investigative Site 208, Yangzhou, Jiangsu
  - Connect Investigative Site 212, Changchun, Jilin
  - Connect Investigative Site 220, Shenyang, Liaoning
  - Connect Investigative Site 207, Shanghai, Shanghai Municipality
  - Connect Investigative Site 218, Shanghai, Shanghai Municipality
  - Connect Investigative Site 221, Taiyuan, Shanxi
  - Connect Investigative Site 222, Taiyuan, Shanxi
  - Connect Investigative Site 224, Ürümqi, Xinjiang
  - Connect Investigative Site 217, Ningbo, Zhejiang
- Hungary (2):
  - Connect Investigative Site 304, Püspökladány, Hajdú-Bihar
  - Connect Investigative Site 303, Szombathely, Vas County
- Poland (9):
  - Connect Investigative Site 402, Krakow, Lesser Poland Voivodeship
  - Connect Investigative Site 401, Krakow, Lesser Poland Voivodeship
  - Connect Investigative Site 403, Lubin, Lower Silesian Voivodeship
  - Connect Investigative Site 408, Wroclaw, Lower Silesian Voivodeship
  - Connect Investigative Site 406, Skierniewice, Lódzkie
  - Connect Investigative Site 404, Bialystok, Podlaskie Voivodeship
  - Connect Investigative Site 405, Bialystok, Podlaskie Voivodeship
  - Connect Investigative Site 410, Częstochowa, Świętokrzyskie Voivodeship
  - Connect Investigative Site 407, Skarżysko-Kamienna, Świętokrzyskie Voivodeship
- South Korea (4):
  - Connect Investigative Site 505, Incheon, Gyeonggi-do
  - Connect Investigative Site 503, Seongnam-si, Gyeonggi-do
  - Connect Investigative Site 501, Seoul, Seoul Teugbyeolsi
  - Connect Investigative Site 502, Seoul, Seoul Teugbyeolsi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kerwin E, Yang T, Su N, Guo J, Adivikolanu R, Longphre M, Wang J, Yun J, Pan W, Wei Z, Collazo R. Rademikibart Treatment for Moderate-to-Severe Uncontrolled Asthma: A Phase 2B Randomized Clinical Trial. Am J Respir Crit Care Med. 2025 May;211(5):749-758. doi: 10.1164/rccm.202409-1708OC. PMID 39998473